CLINICAL TRIAL: NCT03357302
Title: Risk Factors Associated With the Global Burden of Disease in Reunion Island and Comparison With Mainland France and Indian Ocean Countries
Acronym: AVIRON-2
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/CHU/15
Record Dates: First submitted 2017-11-24; First posted 2017-11-29 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Disability or Chronic Disease Leading to Disablement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The question posed by this project is that of the regional estimate of the relative importance of the risk factors of the main pathologies. Our hypothesis is that these risk factors are of different relative importance in Reunion Island compared to metropolitan France.

DETAILED DESCRIPTION:
The definition of health priorities in a given territory is a major field of Public Health research. The World Health Organization has been conducting the Global Burden of Disease study since the 1990s. This study, which has been the subject of numerous publications, aims at estimating the burden for a given population of different causes of mortality and morbidity. It defines a standardized measure allowing comparisons between different countries. The measure developed internationally is the "Disability-adjusted life year" (DALY). This also allows the monitoring of the relative importance of each pathology. This standardized classification of the relative importance of the pathologies and risk factors involved is a major public health tool.

This measure was developed at the international level initially and then recently applied locally (London neighborhoods, US states). For the Indian Ocean zone, DALY values are available for Madagascar, Seychelles and Mauritius. The estimate of this measure for Reunion Island is based on data from metropolitan France. It therefore uses for Reunion mortality, morbidity, income per capita and social indicators of metropolitan France. It does not take into account the specificities of Reunion. In order to better understand Reunion's public health priorities, it seems important to decline this measure at the regional level. The implementation of this measure at the regional level corresponds to the research project AVIRON which aimed at collecting all the data for the calculation of the DALY in Reunion Island. The AVIRON-2 study, which extends AVIRON's focus on morbidity and mortality, will aim at determining the attributable part of the various disease risk factors and to classify these risk factors according to their importance in a given population for all diseases.

ELIGIBILITY:
Inclusion Criteria:

The whole population living in Reunion Island

Exclusion Criteria:

People not living in Reunion Island

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population living in Reunion Island
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Quantity of DALY lost for each risk factor | 2 months after legal and ethical agreements
  Risk factors associated to the most prevalent diseases

CONTACTS AND LOCATIONS:
Overall Officials: Laetitia Huiart, MD, Study Director — Luxembourg Institute of Health
Locations (1):
- Olivier MAILLARD, Saint-Pierre, Reunion, France

IPD SHARING:
Plan to Share IPD: No